CLINICAL TRIAL: NCT03654365
Title: Once Lifetime Hepatitis C (HCV) Screening Among Adults Using Advanced Electronic Population Health Tools and Personal Health Record Tools Tied to an Advanced Electronic Health Record (EHR).
Brief Title: Advanced Electronic Population Health and Personal Health Record Tools to Improve Once Lifetime Hepatitis C Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, David Kaelber MD, Physician and Chief Medical Informatics Officer, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IRB16-00776
Record Dates: First submitted 2018-06-26; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
Keywords: preventative screening; electronic health records; personal health records; population health tools
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Pts in the control arm receive usual care. Usual care includes a EHR based reminder of single HCV testing for patients who are in the birth cohort. (routine alerting)
  Interventions: Other: Routine alerting
- Intervention (Experimental): Pts in the intervention arm receive bulk messaging and bulk ordering of the HCV ab test.
  Interventions: Other: Bulk ordering and bulk messaging; Other: Routine alerting

INTERVENTIONS:
Other: Bulk ordering and bulk messaging — Patients in the intervention group had the hepatitis screening test ordered for them in bulk and then a bulk message sent to them through the personal health record describing hepatitis C and how they could be tested.
  Arms: Intervention
Other: Routine alerting — Passive alerting to providers (during face-to-face encounters using the electronic health record) and to patient (when they review preventative screening recommendations through their personal health record).

SUMMARY:
This study involves randomizing patients due for once in a lifetime Hepatitis C screening based on Center for Disease Control and Prevention and United States Preventative Services Task Force guidelines in one of three primary care clinics within the MetroHealth System to bulk messaging and bulk ordering for HCV antibody vs usual care (routine alerting).

DETAILED DESCRIPTION:
All patients had to have an active personal health record account at the time of being randomized.

Patients had to have been seen by their primary care provider in the last 6 months to be eligible and therefore had a "missed opportunity" for Hepatitis C screening.

Control group received "usual care" which in our system included alert (health maintenance reminder) to the primary care provider at the time of the visit and passive alert in their personal health record (i.e. an alert if they log into their personal health record and look for reminders for preventative care that it due/overdue).

Intervention group received same care as control group plus automatic ordering of the hepatitis C screening test and active electronic letter their personal health record that they were due for hepatitis C screening, what hepatitis C is, what the testing and if positive, treatment could involve, and instruction to go to one of the laboratories in the healthcare system to have their blood drawn if they were interested in the testing.

ELIGIBILITY:
Inclusion Criteria:

* seen recently in one of the three primary care study sites and have an active person health record at the time of randomization; and meet Centers for Disease Control and Prevention/United States Preventative Services Task Force guidelines for once in a lifetime hepatitis C screening

Exclusion Criteria:

* already had once in a lifetime screen for hepatitis C or positive for hepatitis C (by lab test or International Classification of Disease code)

Ages: 51 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-03-25 (Actual)

PRIMARY OUTCOMES:
Impact on hepatitis C antibody testing rates at 12 weeks post direct patient messaging | 12 weeks post-intervention
  Number of patients who remain untested for HCV at 12 weeks post direct patient messaging

SECONDARY OUTCOMES:
Impact of bulk ordering vs bulk messaging and bulk ordering on HCV antibody testing rates | 12 weeks post-intervention
  Assessment of if the patient in the intervention group seemed have the hepatitis screening done just because they were having other blood work done versus specifically wanting to be screened for hepatitis C.